CLINICAL TRIAL: NCT04604574
Title: Evaluating the Integration of Indigenous Healing With Principals of Seeking Safety for Treatment of Indigenous Patients With a History of Trauma and Active Substance Use Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Sciences North Research Institute (Other)
Collaborators: North Shore Tribal Council (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 6010991
Record Dates: First submitted 2020-10-13; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Substance Use Disorders; Post-Traumatic Stress Disorder; Intergenerational Trauma
Keywords: Indigenous Health; Seeking Safety; Health Care Utilization; Residential Addiction Treatment
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Historical Trauma; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: We plan to conduct a pre/post intervention matched comparison group study. We will compare historical treatment outcomes for past Benbowopka patients to outcomes following IHSS treatment for Indigenous patients with a history of trauma and SUD. All patient data will be anonymized at the time of data entry. Propensity matching will be undertaken for patient characteristics, including sex/gender, age, and substance use type. The National Native Alcohol and Drug Abuse Program (NNADAP) tool will be used to analyze the program objective; that is, whether completion rates improve following the implementation of the IHSS intervention. Additionally, a Client Quality Assurance Survey (attached) will be utilized to determine patient satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre/Post-Intervention (Other): Patients who receive the novel IHSS intervention will be compared to historical controls who received the abstinence-based treatment model.
  Interventions: Other: Indigenous Healing and Seeking Safety

INTERVENTIONS:
Other: Indigenous Healing and Seeking Safety — Indigenous Healing and Seeking Safety Intervention: Initial 90-minute meetings will be conducted with the participants; during these meetings, participants will receive information about IHSS, traditional healing, sharing circles, sweat lodge ceremonies, and program details. The sharing circles will take place at Benbowopka Residential treatment Centre in Blind River, Ontario. Each of the sharing circles will be cofacilitated by two Indigenous health-care workers. These facilitators will organize and lead sharing circles daily throughout the 28-day treatment cycle. Each sharing circle will be two hours long. The Seeking Safety program consists of up to 25 treatment topics that aim to teach participants a variety of skills. The majority of topics address the cognitive, behavioral, interpersonal, and case management needs of persons with SUD and posttraumatic stress disorders (PTSD) (Najavits, 2002a). The treatment will adhere to the concept of Two-Eyed Seeing and cultural sensitivity.
  Other Names: Abstinence-Based Treatment Historical Control

SUMMARY:
Background: The negative health outcomes experienced by Indigenous peoples may be understood as direct consequences of colonization. One of the key consequences of the colonial influence on Canada's Indigenous peoples has been intergenerational trauma (IGT). Indigenous communities in Canada face significant challenges with IGT, which often manifest in substance use disorders (SUD). Indigenous communities have identified SUD as one of their greatest health challenges(Maté 2009), with some Northern Ontario First Nations communities experiencing SUD rates of 70% (Calveson 2010). Most Elders, traditional healers, and Indigenous scholars agree that connecting treatment to culture, land, community, and spiritual practices is a pathway to healing trauma and SUD for Indigenous peoples. Recent work by Dr. Teresa Naseba Marsh has demonstrated that Indigenous Healing and Seeking Safety (IHSS) model for trauma therapy can be effectively combined for the treatment of Indigenous patients with a history of trauma and SUD. Seeking Safety incorporates the inclusion of the mind, body, spirit, and self-awareness during treatment, and the perspective of Seeking Safety is convergent with traditional Indigenous healing methods. Benbowopka Treatment Centre is a residential treatment site operated by Mamaweswen, located in the North Shore Tribal Council in Blind River, Ontario. Benbowopka's mandate is to provide treatment for Indigenous clients with trauma and SUD. They are also implementing a culturally sensitive program grounded in IHSS methodology for the treatment of Indigenous patients' trauma and SUD. Through our current collaboration with Benbowopka and Mamaweswen the applicants have collected baseline data from client files to establish historical outcomes going back three years. In 2016, we began the collaborative implementation of the Indigenous Healing and Seeking Safety (IHSS) model for trauma therapy for clients at Benbowopka.

Objective: The purpose of this proposal is to evaluate the effectiveness of the IHSS intervention which blends Indigenous Healing Practices and a mainstream treatment model, Seeking Safety for the treatment of Indigenous patients with a history of trauma and SUD. Methodology: In collaboration with the North Shore Tribal Council and the Benbowopka Treatment Center, we propose a prospective evaluation of IHSS treatment for Indigenous patients with a history of trauma and SUD. Benbowopka treats approximately 90 patients per year in a residential treatment program, and the program has high quality retrospective data on their programming and outcomes. We propose to benchmark anonymized historical program outcomes by evaluating program outcomes and the impact of program completion on health systems usage. Impact of treatment on health system usage will be determined by linking anonymized patient records with records at the Institute for Clinical and Evaluative Sciences (ICES). ICES linkage will provide further insight into hospitalizations, interaction with emergency, mental health, and primary care usage before and following the implementation of the IHSS intervention. We will respect the Tricouncil Policy Statement, Chapter 9, which highlights the importance of engaging with First Nations throughout all phases of the research process. In addition, we will honour Indigenous knowledge by engaging with Elders and the North Shore Tribal council. Through the data governance protocols established at ICES, we will respect the First Nations principles of ownership, control, access and possession of data (OCAP™). Dr. Jennifer Walker Canada Research Chair in Indigenous Health at the Center for Rural and Northern Health Research and ICES Scientist will oversee the process of data sharing and linking de-identified Benbowopka treatment data to anonymized health system data at ICES. Benbowopka and the North Shore Tribal council will maintain complete ownership over the study data and its subsequent dissemination. Anticipated Outcome: We expect that patients who are treated in the IHSS treatment model will have improved outcomes as compared to previous patients of Benbowopka treated under the abstinence based model of therapy. Objectives measures will include treatment completion, substance use at program completion, substance use at follow-up, ED visits, hospitalization, and death. Patient satisfaction will be tracked using surveys administered at treatment completion and is expected to improve with implementation of IHSS. Impact: We expect to demonstrate that the IHSS is a culturally sensitive and effective treatment model for Indigenous patients who are affected by trauma and substance use disorder.

DETAILED DESCRIPTION:
Background:

Indigenous Ways of Knowing coupled with Indigenous Healing provide the foundation for achieving personal and community wellness. Specific health outcomes experienced by Canada's Indigenous Peoples- including trauma and substance use disorders (SUD)-are seen as a direct consequence of colonization. Most notably, these effects are seen in the multi-generational trauma of the residential school system (Kirmayer, et al., 2009; Menzies, 2014; Thatcher, 2004; Stewart, 2008). The aspiration of healing and wellness is most effectively achieved by using tools and methods that are both appropriate and effective for Indigenous Peoples and communities. The evidence suggests that one of the key consequences of the colonial influence on Canada's Indigenous Peoples has been intergenerational trauma, and high rates of depression, suicide, and SUD (Bombay, Matheson, & Anisman, 2009; Kirmayer, et al., 2000; Haskell & Randall, 2009). Intergenerational trauma is the most common term used to describe the systematic trauma suffered by Indigenous Peoples (Evans-Campbell, 2008; Haskell, 2009; Palacios & Portillo, 2009). Intergenerational trauma is now seen as a precursor to depression, anxiety, post-traumatic stress disorder, re-enactment of trauma, suicide, and SUD (Brave Heart, 2004; Duran, 2006; Menzies, 2014; Thatcher, 2004; Waldram, 2006). Indigenous communities in Canada face significant challenges with intergenerational trauma, which often manifest in SUD. Indigenous communities have identified SUD as one of their greatest health challenges, with some Northern Ontario First Nations communities experiencing SUD rates of 70% (Calveson 2010). Between 2004 and 2009, the number of Indigenous patients seeking treatment for SUD in Ontario increased threefold (Calverson 2010). In 2009, the Nishnawbe Aski Nation declared a state of emergency for prescription drug abuse (Prescription Drug Backgrounder; NAN, 2009), and the number of people seeking treatment continues to rise. Many Elders, traditional healers, and Indigenous scholars agree that connecting treatment to culture, land, community, and spiritual practices is a pathway to healing trauma and SUD for Indigenous Peoples. To address SUD for Indigenous patients, Mamaweswen, The North Shore Tribal Council operate the Benbowopka Treatment Centre. Benbowopka is a residential treatment site in Blind River, Ontario with a mandate to provide treatment for Indigenous patients with trauma and SUD. Historically, the treatment program at Benbowopka merged Indigenous Healing with an abstinence-based residential treatment model. However, a 2015 program review identified the need to modernize the program to address the increasing number of patients with concurrent trauma and SUD. The skills required to heal from intergenerational trauma and subsequent recovery of identity can be enhanced by cultural practices, Indigenous Healing, the presence of Elders, and through traditional ceremony (Duran, 2006; Menzies, 2014; Thatcher, 2004; Waldram, 2006). Similarly, Seeking Safety (SS) is a validated, manualized psycho-educational counseling program that targets the unique problems resulting from SUD and trauma (Najavits, 2009). Importantly, the perspective of SS is convergent with traditional Indigenous Healing methods. Because of the content and delivery method of SS, the program complements traditional teachings such as holism, relational connection, spirituality, cultural presence, honesty, and respect (Gone, 2008; Lavallée, 2008; Menzies, 2014; Marsh et al., 2016). Benbowopka staff work with the Client's Circle of Care Team to develop the necessary support services to address the client's physical, mental health/addictions and cultural needs as part of their aftercare services once discharged. In 2016, Benbowopka worked with Dr. Teresa Marsh to integrate and implement SS into a novel treatment intervention, known as Indigenous Healing and Seeking Safety (IHSS) (Marsh et al., 2015; Marsh et al., 2016a; Marsh et al., 2016b). The IHSS intervention aims to increase the coping skills of participants and reduce the chance of relapse by emphasizing values such as respect, care, integration, and healing of self (Najavits, 2007). This community-led initiative-with a novel IHSS clinical treatment framework-presents a unique opportunity to study innovative approaches to Indigenous wellness.

Indigenous Healing and Seeking Safety (IHSS) Intervention: Initial 90-minute meetings will be conducted with the participants; during these meetings, participants will receive information about IHSS, traditional healing, sharing circles, sweat lodge ceremonies, and program details. The sharing circles will take place at Benbowopka Residential treatment Centre in Blind River, Ontario. Each of the sharing circles will be cofacilitated by two Indigenous health-care workers. These facilitators will organize and lead sharing circles daily throughout the 28-day treatment cycle. Each sharing circle will be two hours long. The Seeking Safety program consists of up to 25 treatment topics that aim to teach participants a variety of skills. The majority of topics address the cognitive, behavioral, interpersonal, and case management needs of persons with SUD and posttraumatic stress disorders (PTSD) (Najavits, 2002a). To adhere to the concept of Two-Eyed Seeing and cultural sensitivity, the material will be conveyed verbally. The facilitators will encourage a language that respects the participants' cultural values and beliefs. To encourage a holistic view of mental health and substance use (which includes connection to community), Indigenous healing practices will be incorporated into the sharing circles. Each sharing circle will be opened and closed with smudging, ceremonial drumming, and singing. Tobacco-a herb recognized in Indigenous culture for its healing powers-will be prepared in bundles in advance of the sharing circles. It will be offered to each participant for protection and healing. The cultural coordinator and facilitators will introduce their sacred items and sacred bundle during the sharing circles. A sacred bundle can consist of one or many items. It can be a tobacco or sacred medicine pouch worn around the neck, or it can be an item such as a sacred pipe that the spirits have given to a person to carry for the people. The sacred bundle is considered a very precious possession that represents a person's spiritual life (Hart, 2010; Menzies, 2010). The participants will be invited to bring their bundles, and will be encouraged to place their sacred bundles or items at the center of the circle. Participants will also partake in at least three sweat lodge ceremonies held once a week during the four-week cycle of the intervention period. Sweat lodge ceremonies will provide a powerful way to bring forth Two-Eyed Seeing as an Indigenous decolonizing methodology. The sweat ceremonies help repair the damage done to the spirits, minds, and bodies of the participants. During the sweat ceremonies, the cultural coordinator will give teachings about Aboriginal traditional healing and its restorative power. Participants will also be invited to share their stories and experiences. Also, participants will attend at least two Sacred Fire ceremonies with the staff and cultural coordinator with the purpose of helping them let go of past traumas and substances. Mamaweswen North Shore Community Health Services currently provides a range of physical and mental health/addictions pre-treatment and aftercare services to the seven Member First Nation communities in our area. Each First Nation community in our area also provides some pre-treatment and aftercare services. All of these services work closely with Benbowopka Treatment Centre around the referral and transitioning of clients between required mental health and addiction services. Mamaweswen North Shore Community Health Services has continued on with its community opiate withdrawal program on Sagamok Anishnawbek and has now established an additional partnership with the Sault Ste. Marie Indian Friendship Centre to offer community opiate withdrawal to First Nation individuals who are living in Sault Ste. Marie.

Objective: This proposal aims to evaluate the effectiveness of the treatment model Indigenous Healing and Seeking Safety (IHSS) for the treatment of Indigenous patients with a history of trauma and SUD. Study findings will be used to inform trauma and SUD residential treatment programming and implementation for Indigenous communities across Canada. Our work will contribute to the field of community-based trauma and addiction programming by addressing objectives that consider:

i) the patient perspective; does patient satisfaction improve when IHSS methodology for treatment of trauma and SUD replaces an abstinence-focused approach? ii) the program perspective; do program completion rates improve following the implementation of IHSS intervention? iii) the community perspective; do health system outcomes in the year following treatment completion decrease following IHSS implementation?

Hypothesis: We expect that patients who are treated with the IHSS model will have improved treatment satisfaction (increase of 10% over pre-intervention rates), improved treatment completion (increase of 10% over pre-intervention rates), and a greater reduction in health system usage for addiction-related services at one-year follow-up compared to those treated within the abstinence-based model (decrease of 10% over preintervention rates).

Community Partnership:

The Mamaweswen (North Shore Tribal Council) and the Benbowopka Treatment Centre represent seven member communities (Batchewana, Garden River, Thessalon, Sagamok, Mississauga, Atikameksheng, and Serpent River) on the North Shore of Lake Huron. Mamaweswen and our research group began collaborating on the evaluation of the IHSS protocol in the fall of 2016. The primary research questions and the research approach were developed and supported at the community level. Improving care for community members who are affected by trauma and SUD is a priority for Mamaweswen, the North Shore Tribal Council; it is also a shared research interest with collaborators from the Northern Ontario School of Medicine (NOSM) and the Institute for Clinical and Evaluative Sciences (ICES). Together, Mamaweswen, NOSM, and ICES are aiming to build reciprocal capacity building processes that enable academic collaborators to understand the context of community priorities and allow the community to build capacity for future research and quality improvement initiatives.

Benbowopka Treatment Centre employs a culturally-based residential substance use treatment program, following the Seven Grandfather Teachings. Through these Aboriginal teachings and principles, individuals will learn to understand and accept that they are out of balance-according to the Medicine Wheel-as a result of their SUD. As patients move along the road to recovery, they will learn how to maintain balance and harmony in their mental, physical, emotional, and spiritual health. Individuals will participate in individual counselling, group educational sessions, and talking circles; they will also learn relaxation techniques (through yoga and drumming), the importance of addressing their physical health through proper nutrition and exercise, and how to address their spiritual health through cultural activities and teachings. Benbowopka also endorses medication-assisted treatment with buprenorphine/naloxone for patients with opioid use disorder.

The Northern Ontario School of Medicine (NOSM) is a made-in-the-North medical school that has an innovative model of community-engaged medical education and research, while staying true to its social accountability mandate of improving the health of the people and communities of Northern Ontario. NOSM brings together over 90 community partners, over 1,400 clinical, human, and medical sciences faculty, and more than 200 employees. NOSM's success is very much a result of partnerships and collaborations with individuals, communities, and organizations, including Indigenous communities. The Institute for Clinical and Evaluative Sciences (ICES) is a not-for-profit research institute encompassing a community of research and clinical experts, and a secure and accessible array of Ontario's health-related data. ICES has a special focus to enhance the health of Indigenous peoples through a collaboration with the Chiefs of Ontario.

Methodology:

Design: We plan to conduct a pre/post intervention matched comparison group study. We will compare historical treatment outcomes for past Benbowopka patients to outcomes following IHSS treatment for Indigenous patients with a history of trauma and SUD. All patient data will be anonymized at the time of data entry. Propensity matching will be undertaken for patient characteristics, including sex/gender, age, and substance use type. The National Native Alcohol and Drug Abuse Program (NNADAP) tool will be used to analyze the program objective; that is, whether completion rates improve following the implementation of the IHSS intervention. Additionally, a Client Quality Assurance Survey will be utilized to determine patient satisfaction.

Sample and Study Window: The pre-IHSS intervention study window will span the 36 months prior to the implementation of the IHSS intervention (April 1, 2013 - March 31, 2016; n=343), and the Post-IHSS intervention study window will span the 27 months post-IHSS implementation (January 1, 2018 - March 31, 2020; n>300). We will only include data from patients initiating treatment at Benbowopka during the study window. Patient follow-up will occur in the one year following treatment completion and/or discontinuation. Anonymized patient records will be linked via Ontario Health Insurance Plan (OHIP) number, or Indian Registry Number, to the administrative health data at the ICES, and we will query data in the one year following completion or discontinuation of IHSS at Benbowopka to ascertain impact of substance use on health outcomes including hospitalization, ED visits and opioid-related overdose. For patients with multiple admissions, the date of first admission will serve as the index date for health outcomes evaluation. Treatment Setting: Benbowopka treats approximately 100 patients per year in a residential treatment program, and the program has high quality retrospective data based on standardized assessment screening tools routinely used by the Drug and Alcohol Treatment Information System and the National Native Alcohol and Drug Abuse Program. For the 343 patients admitted between April 1, 2013 and March 31, 2016 86% were Indigenous, 57% male, 84% had alcohol as the primary substance and 38% had opioids as the primary or secondary substance with 65% of patients completing the program.

Access to Linked Administrative Health Data: We propose to link de-identified patient data to record-level provincial health systems data at ICES. ICES routinely links partner data to its core health systems data holdings. ICES linkage will enable virtual follow-up of Benbowopka patients for health systems usage. The main data required for this analysis are available at ICES.

Data Governance: We will respect the Tri-council Policy Statement, Chapter 9, which highlights the importance of engaging with First Nations throughout all phases of the research process. In addition, we will honour Indigenous knowledge by engaging with Elders and the Mamaweswen Council. Anonymized data collected at Benbowopka will be linked in accordance with data governance protocols and data-linkage process established at ICES in consultation with the Chiefs of Ontario. All parties involved in the study will respect Indigenous principles of OCAP.

Planned Analysis:

Using anonymized Benbowopka/ICES-linked data, we propose to evaluate the pre/post-IHSS intervention outcomes. This analysis strategy will provide insight into i) patient satisfaction, ii) program completion, iii) and health systems outcomes for Benbowopka patients. A detailed schematic of the analysis plan is provided in adjacent figure. Baseline metrics will be established for April 1 2013 - March 31 2016 (n = 343) and will be compared to January 1 2018 - March 31, 2020 (n>300) with a one year follow up for health systems outcomes. Specific variables to address patient wellbeing will be captured in the patient satisfaction survey and structures assessments at patient enrollment. Anonymized linked data outcomes from ICES will include primary care visits, mental health visits, initiation of opioid agonist therapy, ED visits, hospitalizations, and all cause mortality.

Training:

Wellness, training, and capacity building are cornerstones to the application. Clinicians at Benbowopka have been trained in the IHSS methodology (beginning January 2016), and IHSS is now routinely delivered to patients. The investigators have worked with Benbowopka team to digitize the data collection and maintenance of their health record system. Establishing a digital health record has enabled efficient data capture and evaluation for quality improvement, research, and reporting purposes. Benbowopka staff, patients, and the Mamawesen communities will benefit from this training and technology enhancement going forward. Importantly, the reciprocal training and skills developed by the community and research team will strongly position collaboration for future community-based research studies, and it will materially increase the capacity for high-quality Indigenous Wellness research in Northern Ontario. Community-based trainees will include three clinical staff, a community-based graduate student, and a research assistant based in the community. The academic research team will also benefit from enhancing its understanding of Indigenous Healing, unique community perspectives, and Indigenous ways of knowing.

Anticipated Outcome:

We will evaluate the results of the IHSS intervention against three distinct primary outcomes. The lens applied to these outcomes will consider:

i) the patient perspective; we will use Client Quality Assurance Survey tool to assess the appropriateness and satisfaction of the intervention ii) the program perspective; we will use the structured assessments at admission to characterize changes in the patient population and the program completion rate as primary outcome to assess the effectiveness of the IHSS intervention iii) the community perspective; we will use the change in substance use related health system usage between the year prior and the year following treatment completion as an indication of the impact of the admission on health system outcomes. We believe our study findings may validate an innovative approach for effective and appropriate care for patients with intergenerational trauma and SUD. We expect that patients who are treated in the IHSS treatment model will have improved satisfaction and outcomes as compared to previous patients of Benbowopka who were treated under the abstinence based model of therapy. Objective measures will include pattern of substance use at admission (to characterize changes in the patient population), treatment completion, and reduction in health system outcomes in the year following treatment compared to the year prior to admission.

Impact and Knowledge Translation:

A material benefit for the community partners will be the digitization of data collection process. For Benbowopka, digitization will enable enhanced ease of program evaluation, reporting, and future quality improvement and research initiatives. Outcomes of the proposed collaboration will use a push, pull, and exchange strategy to benefit the Mamaweswen, Benbowopka, and stakeholders who have an interest in programming and implementation of trauma and SUD treatment.

Push Strategy: Collaboratively, we will actively disseminate the study findings to stakeholders, including Indigenous Health Authorities, Provincial and Federal funding agencies, and community-based treatment programs. Specifically, we will organize in-person presentations to the Chiefs of Ontario and Mamaweswen North Shore Tribal Council. Data will be provided to stakeholders via print, digital, and social media (Facebook/Twitter) via presentation, infographic and explainer video format.

Pull Strategy: We also propose to make study findings freely available on the Benbowopka, Mamaweswen, and other partner websites. Detailed study findings may also be made available via open source peer-reviewed publication. Social media hashtags and user groups will target those who may wish to 'pull' the freely available study findings.

Exchange: To ensure that the necessary knowledge users are directly engaged, a multidisciplinary team of stakeholders will be assembled for in-person meetings and webinars to discuss study outcomes and recommendations for planning and implementation. These stakeholders will include community members, leaders in the field of Indigenous Health, provincial and federal healthcare funders, and academic researchers. In addition to internet-based knowledge translation, we will also organize a series of in-person presentations for communities who are served by Benbowopka.

ELIGIBILITY:
Inclusion Criteria:

* Substance Use Disorder
* Intergenerational Trauma

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
the patient perspective | 28 days
  we will use Client Quality Assurance Survey tool to assess the appropriateness and satisfaction of the intervention.
the program perspective | 28 days
  we will use the structured assessments at admission to characterize changes in the patient population and the program completion rate as primary outcome to assess the effectiveness of the IHSS intervention
the community perspective | One Year
  Change in substance use related health system usage (number of Emergency room presentation and number of acute care admissions for substance use related conditions) between the year prior and the year following treatment completion as an indication of the impact of the admission on health system outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David C Marsh, MD, Principal Investigator — Northern Ontario School of Medicine
Locations (1):
- Northern Ontario School of Medicine, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morin KA, Marsh TN, Eshakakogan C, Eibl JK, Spence M, Gauthier G, Walker JD, Sayers D, Ozawanimke A, Bissaillion B, Marsh DC. Community trial evaluating the integration of Indigenous healing practices and a harm reduction approach with principles of seeking safety in an Indigenous residential treatment program in northern Ontario. BMC Health Serv Res. 2022 Aug 16;22(1):1045. doi: 10.1186/s12913-022-08406-3. PMID 35974328